CLINICAL TRIAL: NCT01526057
Title: A RANDOMIZED, DOUBLE-BLIND, STUDY COMPARING THE PHARMACOKINETICS AND PHARMACODYNAMICS, AND ASSESSING THE SAFETY OF PF-05280586 AND RITUXIMAB IN SUBJECTS WITH ACTIVE RHEUMATOID ARTHRITIS ON A BACKGROUND OF METHOTREXATE WHO HAVE HAD AN INADEQUATE RESPONSE TO ONE OR MORE TNF ANTAGONIST THERAPIES
Brief Title: A Pharmacokinetic/Pharmacodynamic Study Comparing PF-05280586 To Rituximab In Subjects With Active Rheumatoid Arthritis With An Inadequate Response To TNF Inhibitors (REFLECTIONS B328-01)
Acronym: REFLECTIONS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B3281001; ICON 9002/010; 2011-002896-40 (EudraCT Number)
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Results first posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-10

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; rituximab; methotrexate; anti-TNF
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A - PF-05280586 (Experimental)
  Interventions: Biological: PF-05280586
- B - Rituximab EU (Active Comparator)
  Interventions: Biological: MabThera
- C- Rituximab-US (Active Comparator)
  Interventions: Biological: Rituxan

INTERVENTIONS:
Biological: PF-05280586 — 1000 mg, IV on days 1 and 15
  Arms: A - PF-05280586
Biological: MabThera — 1000 mg, IV on days 1 and 15
  Arms: B - Rituximab EU
Biological: Rituxan — 1000 mg, IV on days 1 and 15
  Arms: C- Rituximab-US

SUMMARY:
In this study, patients with moderate to severe rheumatoid arthritis who are being treated with methotrexate will receive 2 intravenous treatments with either PF-05280586 or Rituxan (Rituximab) or MabThera (Rituximab). During the course of the study, the effects of the drugs will be assessed by sampling the levels of drug in the blood, blood cell counts, and by comparing these levels among the different treatments. Safety, tolerability and immunologic response also will be evaluated throughout.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of rheumatoid arthritis
* Meets Class I, II or III of the ACR 1991 Revised Criteria
* RA seropositivity
* Stable dose of methotrexate
* Inadequate response to TNF inhibitors

Exclusion Criteria:

* Any prior treatment with lymphocyte depleting therapies
* History of active TB infection
* Known or screen test positive for specific viruses or indicators of viral infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2012-03-20 (Actual); Primary Completion 2013-08-13 (Actual); Study Completion 2014-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (84):
- United States (43):
  - University of Alabama at Bermingham, Birmingham, Alabama
  - University of Alabama at Birmingham - Arthritis Clinical Intervention Program (ACIP) SRC 076, Birmingham, Alabama
  - Rheumatology Associates of North Alabama, PC, Huntsville, Alabama
  - ArthroCare, Arthritis Care & Research, PC, Gilbert, Arizona
  - Mercy Clinic Hot Springs Communities, Hot Springs, Arkansas
  - UCLA David Geffen School of Medicine, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Desert Medical Advances, Palm Desert, California
  - Advances In Medicine, Rancho Mirage, California
  - New England Research Assoc. LLC, Trumbull, Connecticut
  - Arthritis Associates, Orlando, Florida
  - University of South Florida - College of Medicine, Frank and Carol Morsani Center, Tampa, Florida
  - Loyola Center for Health at Burr Ridge, Burr Ridge, Illinois
  - Loyola Medical Medical Center Outpatient Center, Maywood, Illinois
  - Loyola University Medical Center Pharmacy, Maywood, Illinois
  - Illinois Bone and Joint Institute, Morton Grove, Illinois
  - Loyola Center for health at Oakbrook Terrace North, Oakbrook Terrace, Illinois
  - Bluegrass Community Research, Inc., Lexington, Kentucky
  - Klein & Associates, M.D., P.A., Cumberland, Maryland
  - Klein & Associates, M.D., P.A., Hagerstown, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - UMass Memorial Medical Center - Memorial Campus, Worcester, Massachusetts
  - UMass Memorial Medical Center-Rheumatology Center-Memorial Campus, Worcester, Massachusetts
  - Bronson Internal Medicine & Rheumatology, Battle Creek, Michigan
  - Rheumatology/Arthritis Center, Lansing, Michigan
  - University Of Nevada School Of Medicine, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - North Shore-LIJ Health System - Division of Rheumatology and Allergy-Clinical Immunology, Great Neck, New York
  - Box Arthritis & Rheumatology of the Carolinas, PLLC, Charlotte, North Carolina
  - Hickory Family Practice Associates, Hickory, North Carolina
  - PMG Research of Hickory, LLC - PI's Main Office (Subject visit, IP Storage, Infusion, & Lab Draws), Hickory, North Carolina
  - PMG Research of Hickory, Hickory, North Carolina
  - Cincinnati Rheumatic Disease Study Group, Inc., Cincinnati, Ohio
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - The Arthritis Group, Philadelphia, Pennsylvania
  - Clinical Research Center of Reading, LLP, Wyomissing, Pennsylvania
  - Arthritis Associates, PLLC, Hixson, Tennessee
  - Arthritis Clinic, Jackson, Tennessee
  - West Tennessee Research Institute, Jackson, Tennessee
  - Metroplex Clinical Research Center, Dallas, Texas
  - Center For Clinical Trials Of Houston, Houston, Texas
  - Southwest Rheumatology Research LLC., Mesquite, Texas
- Australia (3):
  - Rheumatology Research Unit, Maroochydore, Queensland
  - The Queen Elizabeth Hospital, Department of Rheumatology, Woodville South, South Australia
  - St. Vincent's Hospital (Melbourne), Fitzroy, Victoria
- Canada (5):
  - Pharmacie Matte et Petit, Québec, Quebec
  - Centre de Rhumatologie St-Louis, Québec, Quebec
  - Centre de Rhumatologie de l'Est du Quebec, Rimouski, Quebec
  - Clinique Medicale du Phare, Rimouski, Quebec
  - Centre de Recherche Musculo-Squelettique, Trois-Rivières, Quebec
- Colombia (12):
  - Clinica Medellin S.A Sede Centro, Medellín, Antioquia
  - Mix Supplier S.A, Medellín, Antioquia
  - Rodrigo Botero S.A.S., Medellín, Antioquia
  - Cediul S.A., Barranquilla, Atlántico
  - Centro de Reumatologia y Ortopedia, Barranquilla, Atlántico
  - Clinica Bonnadona - Prevenir S.A., Barranquilla, Atlántico
  - Clinica de la Costa Ltdz., Barranquilla, Atlántico
  - IPS Centro Integral de Reumatologia del Cairbe, CIRCARIBE S.A.S., Barranquilla, Atlántico
  - Sabbag Radiologos Ltda., Barranquilla, Atlántico
  - Cerid S.A., Barranquilla, Colombia, Atlántico
  - Congregacion de las Hemanas Franciscanas Misioneras de Maria Auxiliadora - Clinica La Asuncion, Barranquilla, Colombia, Atlántico
  - IPS Clinica General del Norte S.A., Barranquilla, Colombia, Atlántico
- Schlosspark-Klinik GMBH, Internal Medicine II, Berlin, Germany
- The Chaim Sheba Medical Center Department of Internal Medicine B, Ramat Gan, Israel
- Mexico (4):
  - Cliditer, S.A. de C.V., México, D.F.
  - Private Office, Guadalajara, Jalisco
  - Centro De Investigacion Y Atencion Integral Durango CIAID, Durango
  - Centro de Alta Especialidad en Reumatologia e Investigacion del Potosi S.C., San Luis Potosí City
- Russia (8):
  - LLC CDCR "Healthy Joints", Novosibirsk, Novosibirsk Oblast
  - GBUZ City Clinical Hospital #7, Kazan', Tatarstan Republic
  - State Institution of Healthcare "Regional Clinical Hospital for Wars' Veterans", Kemerovo
  - State Budgetary Institution of Healthcare of Nizhegorodskiy Region, Nizhny Novgorod
  - St. Petersburg state Healthcare lnstitution 'Clinical Rheumatology Hospital No25, Saint Petersburg
  - Llc Ava-Peter, Saint Petersburg
  - State Institute of Healthcare Samara Regional Clinical Hospital named after M.I.Kalinin, Samara
  - Regional State Budget Institution of Healthcare "Tomsk Regional Clinical Hospital", Tomsk
- South Africa (2):
  - Panorama Medical Centre, Panorama, CAPE TOWN
  - Dr. Jan Fourie Medical Centre, Dundee, KwaZulu-Natal
- United Kingdom (5):
  - Bexley Wing - St. James's University Hospital, Leeds, UK
  - Pharmacy Department, Leeds General Infirmary, Leeds Teaching Hospitals NHS Trust, Leeds
  - "The University of Leeds,, Leeds
  - Pharmacy Dispensing - Bexley Wing - St. James's University Hospital, Leeds
  - Whipps Cross University Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Williams JH, Hutmacher MM, Zierhut ML, Becker JC, Gumbiner B, Spencer-Green G, Melia LA, Liao KH, Suster M, Yin D, Li R, Meng X. Comparative assessment of clinical response in patients with rheumatoid arthritis between PF-05280586, a proposed rituximab biosimilar, and rituximab. Br J Clin Pharmacol. 2016 Dec;82(6):1568-1579. doi: 10.1111/bcp.13094. Epub 2016 Sep 22. PMID 27530379
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3281001&StudyName=A%20Pharmacokinetic/Pharmacodynamic%20Study%20Comparing%20PF-05280586%20To%20Rituximab%20In%20Subjects%20With%20Active%20Rheumatoid%20Arthritis%20With%20An%20Inadequate%20Res

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multinational, randomized, double-blind, controlled trial in participants with active rheumatoid arthritis (RA) on a background of methotrexate (MTX). The study was conducted at 56 centres in 10 countries. There were a total of 220 participants enrolled in this study.
Groups:
- Rituximab-Pfizer: Participants received intravenous (IV) rituximab (PF-05280586) infusion 1000 milligrams per 500 milliliters (preceded by 100 milligram [mg] methylprednisolone, an antipyretic such as paracetamol, and an antihistamine such as diphenhydramine) on Day 1 and 15 and continued to receive a stable background regimen of methotrexate 10 to 25 mg per week (mg/week) (7.5 mg/week in the event of prior poor tolerance) for up to 25 weeks. Folate supplementation was encouraged according to local standard of care.
- Rituximab-European Union (EU): Participants received IV rituximab (MabThera) infusion 1000 milligrams per 500 milliliters (preceded by 100 mg methylprednisolone, an antipyretic such as paracetamol, and an antihistamine such as diphenhydramine) on Day 1 and 15 and continued to receive a stable background regimen of methotrexate 10 to 25 mg/week (7.5 mg/week in the event of prior poor tolerance) for up to 25 weeks. Folate supplementation was encouraged according to local standard of care.
- Rituximab-US: Participants received IV rituximab (Rituxan) infusion 1000 milligrams per 500 milliliters (preceded by 100 mg methylprednisolone, an antipyretic such as paracetamol, and an antihistamine such as diphenhydramine) on Day 1 and 15 and continued to receive a stable background regimen of methotrexate 10 to 25 mg/week (7.5 mg/week in the event of prior poor tolerance) for up to 25 weeks. Folate supplementation was encouraged according to local standard of care.
Period: Overall Study
Arm/Group | Rituximab-Pfizer | Rituximab-European Union (EU) | Rituximab-US
Started | 73 | 74 | 73
Completed | 64 | 71 | 67
Not Completed | 9 | 3 | 6
Not completed — Withdrawal by Subject | 3 | 2 | 2
Not completed — Adverse Event | 3 | 1 | 1
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Other | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT) population included all participants who were randomized and received at least 1 dose of study treatment.
Groups:
- Rituximab-Pfizer: Participants received IV rituximab (PF-05280586) infusion 1000 milligrams per 500 milliliters (preceded by 100 mg methylprednisolone, an antipyretic such as paracetamol, and an antihistamine such as diphenhydramine) on Day 1 and 15 and continued to receive a stable background regimen of methotrexate 10 to 25 mg/week (7.5 mg/week in the event of prior poor tolerance) for up to 25 weeks. Folate supplementation was encouraged according to local standard of care.
- Rituximab-EU: Participants received IV rituximab (MabThera) infusion 1000 milligrams per 500 milliliters (preceded by 100 mg methylprednisolone, an antipyretic such as paracetamol, and an antihistamine such as diphenhydramine) on Day 1 and 15 and continued to receive a stable background regimen of methotrexate 10 to 25 mg/week (7.5 mg/week in the event of prior poor tolerance) for up to 25 weeks. Folate supplementation was encouraged according to local standard of care.
- Total: Total of all reporting groups
Arm/Group | Rituximab-Pfizer | Rituximab-EU | Rituximab-US | Total
Number analyzed (Participants) | 73 | 74 | 73 | 220
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.9 (11.52) | 54.9 (11.07) | 53.4 (11.87) | 54.4 (11.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 57 | 54 | 170
  Male | 14 | 17 | 19 | 50

OUTCOME MEASURES:

1. Primary Outcome: Maximum Serum Concentration (Cmax) of Rituximab
Description: Cmax is the peak serum concentration of study drug (rituximab) after a dose has been administered.
Time Frame: Predose (Day 1) and 3, 4.25 (immediately before 1st infusion end), 72, 168, 335 (Day 15 within 1.5 hours before 2nd infusion), 337.5, 339.25 (Day 15 immediately before 2nd infusion end), 408, 504, 672, 1344, and 2016 hours after start of 1st infusion
Population: Per protocol (PP) population: all participants who were randomized, received the full doses of the assigned study treatment, and had no major protocol violations that could impact the pharmacokinetic (PK) analysis. Exclusions from the PP population were based on a blinded data review by the Medical Monitor and Clinical Pharmacologist.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Rituximab-Pfizer | Rituximab-EU | Rituximab-US
Number analyzed (Participants) | 68 | 67 | 63
micrograms per milliliter | 453 (153) | 422 (111) | 430 (163)
Statistical Analysis 1: Comparison: Rituximab-Pfizer vs Rituximab-EU; A 90% CI on the estimated difference between 2 treatment groups was constructed using a 1-way analysis of variance (ANOVA) model based on natural log-transformed data. The estimated differences for the log-transformed PK parameters were then transformed to relative ratios of PK parameters by exponentiation; Test type: Equivalence — PK similarity for a given test-to-reference comparison would be demonstrated if the 90% CI for the test-to-reference ratios in Cmax and area under the serum concentration-time curve (AUC) from time 0 extrapolated to infinite time (AUC 0-inf) are within the 80.00% to 125.00% range; Test-to-reference ratio: adjusted means = 105.67, 90% CI 2-sided [96.91 to 115.21] — Rituximab-Pfizer is the numerator
Statistical Analysis 2: Comparison: Rituximab-Pfizer vs Rituximab-US; A 90% CI on the estimated difference between 2 treatment groups was constructed using a 1-way ANOVA model based on natural log-transformed data. The estimated differences for the log-transformed PK parameters were then transformed to relative ratios of PK parameters by exponentiation; Test type: Equivalence — PK similarity for a given test-to-reference comparison would be demonstrated if the 90% CI for the test-to-reference ratios in Cmax and AUC 0-inf are within the 80.00% to 125.00% range; Test-to-reference ratio: adjusted means = 106.62, 90% CI 2-sided [97.65 to 116.41] — Rituximab-Pfizer is the numerator
Statistical Analysis 3: Comparison: Rituximab-EU vs Rituximab-US; [analysis description as in outcome 1, analysis 2]; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Test-to-reference ratio: adjusted means = 100.90, 90% CI 2-sided [92.38 to 110.20] — Rituximab-EU is the numerator

2. Primary Outcome: AUC 0-inf of Rituximab
Description: The AUC 0-inf refers to the concentration in serum of the drug over time. It represents the total drug exposure over time, from time 0 (the point of drug administration) extrapolated to infinity.
Time Frame: as for outcome 1
Population: PP population. "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ug*hr/mL
Arm/Group | Rituximab-Pfizer | Rituximab-EU | Rituximab-US
Number analyzed (Participants) | 68 | 67 | 62
ug*hr/mL | 213000 (90400) | 200000 (74500) | 214000 (95300)
Statistical Analysis 1: Comparison: Rituximab-Pfizer vs Rituximab-EU; [analysis description as in outcome 1, analysis 2]; Test type: Equivalence — PK similarity for a given test-to-reference comparison would be demonstrated if the 90% CI for the test-to-reference ratios in Cmax and AUC0-inf are within the 80.00% to 125.00% range; Test-to-reference ratio: adjusted means = 104.19, 90% CI 2-sided [92.75 to 117.06]
Statistical Analysis 2: Comparison: Rituximab-Pfizer vs Rituximab-US; [analysis description as in outcome 1, analysis 2]; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Test-to-reference ratio: adjusted means = 100.45, 90% CI 2-sided [89.20 to 113.11]
Statistical Analysis 3: Comparison: Rituximab-EU vs Rituximab-US; [analysis description as in outcome 1, analysis 2]; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Test-to-reference ratio: adjusted means = 96.40, 90% CI 2-sided [85.57 to 108.60]

3. Secondary Outcome: Rituximab AUC From Time 0 to 2 Weeks (AUC 0-2wk)
Description: The AUC 0-2wk refers to the concentration in serum of the drug over time. It represents the total drug exposure over time, from time 0 (the point of drug administration) to 2 weeks after drug administration.
Time Frame: as for outcome 1
Population: PP population.
Measure: Mean (Standard Deviation); unit: ug*hr/mL
Arm/Group | Rituximab-Pfizer | Rituximab-EU | Rituximab-US
Number analyzed (Participants) | 68 | 67 | 63
ug*hr/mL | 52100 (18000) | 49600 (14200) | 49200 (15900)
Statistical Analysis 1: Comparison: Rituximab-Pfizer vs Rituximab-EU; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Test-to-reference ratio: adjusted means = 103.74, 90% CI 2-sided [95.10 to 113.12] — Rituximab-Pfizer is the numerator
Statistical Analysis 2: Comparison: Rituximab-Pfizer vs Rituximab-US; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Test-to-reference ratio: adjusted means = 105.56, 90% CI 2-sided [96.64 to 115.30] — Rituximab-Pfizer is the numerator
Statistical Analysis 3: Comparison: Rituximab-EU vs Rituximab-US; A 90% CI on the estimated difference between 2 treatment groups was constructed using a 1-way ANOVA model based on natural log-transformed data; Test type: Superiority; Test-to-reference ratio: adjusted means = 101.76, 90% CI 2-sided [93.13 to 111.18] — Rituximab-EU is the numerator

4. Secondary Outcome: Rituximab AUC From Time 0 to the Time of the Last Quantifiable Concentration (AUC 0-T)
Description: The AUC 0-T refers to the concentration in serum of the drug over time. It represents the total drug exposure over time, from time 0 (the point of drug administration) to the last measured concentration at time T.
Time Frame: as for outcome 1
Population: PP population.
Measure: Mean (Standard Deviation); unit: ug*hr/mL
Arm/Group | Rituximab-Pfizer | Rituximab-EU | Rituximab-US
Number analyzed (Participants) | 68 | 67 | 63
ug*hr/mL | 198000 (79600) | 188000 (64300) | 196000 (78300)
Statistical Analysis 1: Comparison: Rituximab-Pfizer vs Rituximab-EU; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Test-to-reference ratio: adjusted means = 103.36, 90% CI 2-sided [92.81 to 115.12]
Statistical Analysis 2: Comparison: Rituximab-Pfizer vs Rituximab-US; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Test-to-reference ratio: adjusted means = 101.33, 90% CI 2-sided [90.82 to 113.04]
Statistical Analysis 3: Comparison: Rituximab-EU vs Rituximab-US; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Test-to-reference ratio: adjusted means = 98.03, 90% CI 2-sided [87.83 to 109.40]

5. Secondary Outcome: CD19+ B-cell Count AUC From Time 0 to the Last Measurement at Time T (AUC 0-T,B-cell)
Description: The AUC 0-T,B-cell refers to the concentration in serum of B-cells. It represents the total B-cells over time from time 0 (the point of drug administration) to the last measurement taken at time T.
Time Frame: Baseline and Weeks 2, 3, 5, 9, 13, 17, 21 and 25 (EOT)
Population: mITT population. "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: cells*day/mL
Arm/Group | Rituximab-Pfizer | Rituximab-EU | Rituximab-US
Number analyzed (Participants) | 68 | 69 | 67
cells*day/mL | 13312 (13309) | 14304 (13146) | 12496 (13500)

6. Secondary Outcome: Minimum Post-Baseline CD19+ B-cell Count (/uL)
Description: The lowest CD19+ B-cell count measured in a participant's blood post-baseline.
Time Frame: Baseline and Weeks 2, 3, 5, 9, 13, 17, 21 and 25 (EOT)
Population: mITT population. "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Rituximab-Pfizer | Rituximab-EU | Rituximab-US
Number analyzed (Participants) | 68 | 69 | 67
cells/uL | 0.0 (0.28) | 0.0 (0.00) | 0.0 (0.18)

7. Secondary Outcome: Time to Minimum Post-Baseline CD19+ B-cell Count (Weeks)
Description: The amount of time in weeks from baseline to the lowest observed CD19+ B-cell count.
Time Frame: Baseline and Weeks 2, 3, 5, 9, 13, 17, 21 and 25 (EOT)
Population: mITT population. "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Rituximab-Pfizer | Rituximab-EU | Rituximab-US
Number analyzed (Participants) | 68 | 69 | 67
weeks | 1.4 (1.41) | 1.6 (1.68) | 1.5 (1.31)

8. Secondary Outcome: Duration of B-cell Depletion (τB-cell) (Days)
Description: The τB-cell is defined as the time interval over which the B-cell count was <0.3 cells/uL or the detection limit.
Time Frame: Baseline and Weeks 2, 3, 5, 9, 13, 17, 21 and 25 (EOT)
Population: mITT population. "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Rituximab-Pfizer | Rituximab-EU | Rituximab-US
Number analyzed (Participants) | 68 | 69 | 67
days | 126 (41.8) | 123 (38.6) | 120 (40.6)

9. Secondary Outcome: Percentage of Participants With CD19+ B-cell Count Recovery
Description: The percentage of participants with CD19+ B-cell counts which fell to <50% of Baseline value during treatment and which recovered to ≥50% of Baseline value at End of Treatment.
Time Frame: Baseline and Weeks 2, 3, 5, 9, 13, 17, 21 and 25
Population: mITT population. "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab-Pfizer | Rituximab-EU | Rituximab-US
Number analyzed (Participants) | 68 | 69 | 67
Percentage of participants | 4.4 | 8.7 | 9.0

10. Secondary Outcome: Area Under the CD19+ B-cell Count Concentration-time Profile (AUC 0-T, B-cell)
Description: The AUC 0-T, B-cell refers to the CD19+ B-cell count over time. It represents the total B-cells over time, from time 0 (the point of drug administration) to the last measured count at time T.
Time Frame: Baseline and Weeks 2, 3, 5, 9, 13, 17, 21 and 25 (EOT)
Population: mITT population. "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: cells*day/uL
Arm/Group | Rituximab-Pfizer | Rituximab-EU | Rituximab-US
Number analyzed (Participants) | 68 | 69 | 67
cells*day/uL | 13312.1 (13309.15) | 14304.2 (13145.72) | 12495.9 (13499.97)

11. Secondary Outcome: Baseline and Change From Baseline in Circulating Immunoglobulin-M (IgM) by Visit (Grams Per Liter (g/L])
Description: The level of IgM in serum at Baseline and the change from Baseline at each subsequent visit.
Time Frame: Baseline and Weeks 1, 2, 3, 4, 5, 9, 13, 17, 21 and 25 (EOT)
Population: mITT population. "Number Analyzed" = participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Rituximab-Pfizer | Rituximab-EU | Rituximab-US
Number analyzed (Participants) | 73 | 74 | 73
g/L
  Baseline | 1.381 (0.7617) | 1.460 (0.8076) | 1.394 (0.8372)
  Change from Baseline at Week 1: number analyzed (Participants) | 71 | 69 | 70
  Change from Baseline at Week 1 | 0.0 (0.15) | 0.0 (0.17) | -0.0 (0.19)
  Change from Baseline at Week 2: number analyzed (Participants) | 71 | 72 | 68
  Change from Baseline at Week 2 | 0.0 (0.17) | 0.0 (0.17) | 0.0 (0.20)
  Change from Baseline at Week 3: number analyzed (Participants) | 71 | 74 | 69
  Change from Baseline at Week 3 | -0.1 (0.18) | -0.1 (0.17) | -0.0 (0.15)
  Change from Baseline at Week 4: number analyzed (Participants) | 68 | 69 | 68
  Change from Baseline at Week 4 | -0.1 (0.27) | -0.1 (0.20) | -0.0 (0.33)
  Change from Baseline at Week 5: number analyzed (Participants) | 72 | 71 | 69
  Change from Baseline at Week 5 | -0.1 (0.3) | -0.1 (0.26) | -0.1 (0.23)
  Change from Baseline at Week 9: number analyzed (Participants) | 68 | 73 | 70
  Change from Baseline at Week 9 | -0.2 (0.32) | -0.3 (0.27) | -0.2 (0.28)
  Change from Baseline at Week 13: number analyzed (Participants) | 67 | 72 | 67
  Change from Baseline at Week 13 | -0.2 (0.52) | -0.3 (0.30) | -0.2 (0.55)
  Change from Baseline at Week 17: number analyzed (Participants) | 67 | 71 | 67
  Change from Baseline at Week 17 | -0.1 (0.92) | -0.3 (0.34) | -0.3 (0.34)
  Change from Baseline at Week 21: number analyzed (Participants) | 60 | 65 | 60
  Change from Baseline at Week 21 | -0.3 (0.42) | -0.4 (0.33) | -0.3 (0.35)
  Change from Baseline at Week 25: number analyzed (Participants) | 50 | 57 | 55
  Change from Baseline at Week 25 | -0.4 (0.42) | -0.3 (0.30) | -0.3 (0.48)

12. Secondary Outcome: Percent (%) Change From Baseline in Circulating IgM by Visit (g/L)
Description: The percentage change from Baseline in circulating IgM by visit.
Time Frame: Baseline and Weeks 1, 2, 3, 4, 5, 9, 13, 17, 21 and 25
Population: mITT population. "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure. "Number Analyzed" = participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Rituximab-Pfizer | Rituximab-EU | Rituximab-US
Number analyzed (Participants) | 72 | 74 | 70
percent change
  Week 1: number analyzed (Participants) | 71 | 69 | 70
  Week 1 | 3.3 (18.62) | 1.4 (9.57) | -0.5 (9.93)
  Week 2: number analyzed (Participants) | 71 | 72 | 68
  Week 2 | 0.1 (12.45) | -0.3 (9.42) | 0.7 (14.06)
  Week 3: number analyzed (Participants) | 72 | 74 | 69
  Week 3 | -3.4 (12.98) | -4.9 (9.95) | -2.7 (9.82)
  Week 4: number analyzed (Participants) | 68 | 69 | 68
  Week 4 | -5.5 (14.77) | -5.0 (10.59) | -2.2 (21.89)
  Week 5: number analyzed (Participants) | 72 | 71 | 69
  Week 5 | -8.6 (16.00) | -7.9 (15.60) | -5.6 (14.39)
  Week 9: number analyzed (Participants) | 68 | 73 | 70
  Week 9 | -14.4 (13.68) | -16.9 (13.69) | -14.1 (13.73)
  Week 13: number analyzed (Participants) | 67 | 72 | 67
  Week 13 | -11.5 (37.17) | -22.2 (13.92) | -16.2 (30.14)
  Week 17: number analyzed (Participants) | 67 | 71 | 67
  Week 17 | 5.5 (226.39) | -23.7 (16.35) | -21.6 (14.88)
  Week 21: number analyzed (Participants) | 60 | 65 | 60
  Week 21 | -21.6 (17.72) | -24.7 (21.00) | -21.3 (15.69)
  Week 25: number analyzed (Participants) | 50 | 57 | 55
  Week 25 | -24.2 (14.63) | -21.0 (16.95) | -20.5 (21.78)

13. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 20% Improvement (ACR20) Response by Visit
Description: ACR20 response: greater than or equal to (≥)20% improvement in tender joint count; ≥20% improvement in swollen joint count; and ≥20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP).
  Non-responder imputation categorized participants as having a non-response if they did not have data available at a visit due to missing data or study discontinuation. Participants who rolled over to the extension study were not included in the non-responder imputation from that point on.
Time Frame: Weeks 3, 5, 9, 13, 17, 21 and 25
Population: mITT population. "Number Analyzed" = participants evaluable at specified time points.
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab-Pfizer | Rituximab-EU | Rituximab-US
Number analyzed (Participants) | 73 | 74 | 73
Percentage of participants
  Week 3 | 34.2 | 33.8 | 32.9
  Week 5 | 54.8 | 56.8 | 42.5
  Week 9 | 49.3 | 60.8 | 58.9
  Week 13 | 50.7 | 70.3 | 63.0
  Week 17 | 54.8 | 67.6 | 67.1
  Week 21: number analyzed (Participants) | 72 | 74 | 72
  Week 21 | 54.2 | 62.2 | 69.4
  Week 25: number analyzed (Participants) | 62 | 63 | 62
  Week 25 | 50.0 | 60.3 | 71.0

14. Secondary Outcome: Percentage of Participants With ACR 70% Improvement (ACR70) Response by Visit
Description: ACR70 response: ≥70% improvement in tender joint count; ≥70% improvement in swollen joint count; and ≥70% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
  Non-responder imputation categorized participants as having a non-response if they did not have data available at a visit due to missing data or study discontinuation. Participantss who rolled over to the extension study were not included in the non-responder imputation from that point on.
Time Frame: Weeks 3, 5, 9, 13, 17, 21 and 25 (EOT)
Population: mITT population. "Number Analyzed" = participants evaluable at specified time points.
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab-Pfizer | Rituximab-EU | Rituximab-US
Number analyzed (Participants) | 73 | 74 | 73
Percentage of participants
  Week 3 | 2.7 | 2.7 | 2.7
  Week 5 | 6.8 | 6.8 | 8.2
  Week 9 | 12.3 | 17.6 | 16.4
  Week 13 | 19.2 | 28.4 | 20.5
  Week 17 | 15.1 | 18.9 | 19.2
  Week 21: number analyzed (Participants) | 72 | 74 | 72
  Week 21 | 13.9 | 23.0 | 20.8
  Week 25: number analyzed (Participants) | 62 | 63 | 62
  Week 25 | 16.1 | 17.5 | 19.4

15. Secondary Outcome: Percentage of Participants With ACR 50% Improvement (ACR50) Response by Visit
Description: ACR50 response: ≥50% improvement in tender joint count; ≥50% improvement in swollen joint count; and ≥50% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
  Non-responder imputation categorized participants as having a non-response if they did not have data available at a visit due to missing data or study discontinuation. Participants who rolled over to the extension study were not included in the non-responder imputation from that point on.
Time Frame: Weeks 3, 5, 9, 13, 17, 21 and 25
Population: mITT population. "Number Analyzed" = participants evaluable at specified time points.
Measure: Number; unit: Percentage of Participants
Arm/Group | Rituximab-Pfizer | Rituximab-EU | Rituximab-US
Number analyzed (Participants) | 73 | 74 | 73
Percentage of Participants
  Week 3 | 8.2 | 5.4 | 9.6
  Week 5 | 19.2 | 16.2 | 20.5
  Week 9 | 21.9 | 32.4 | 35.6
  Week 13 | 35.6 | 40.5 | 31.5
  Week 17 | 24.7 | 36.5 | 37.0
  Week 21: number analyzed (Participants) | 72 | 74 | 72
  Week 21 | 27.8 | 37.8 | 38.9
  Week 25: number analyzed (Participants) | 62 | 63 | 62
  Week 25 | 21.0 | 38.1 | 33.9

16. Secondary Outcome: Percentage of Participants by Anti-drug Antibody (ADA) Status
Description: Presence of anti-rituximab antibodies in blood. Participants with a positive antibody status at any time during the study were defined as having overall positive antibody status; participants with a negative antibody status throughout the study were defined as having overall negative antibody status.
Time Frame: Days 1 up to Day 169.
Population: mITT population.
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab-Pfizer | Rituximab-EU | Rituximab-US
Number analyzed (Participants) | 73 | 74 | 73
Percentage of participants | 9.6 | 13.5 | 12.3

17. Secondary Outcome: Percentage of Participants With Neutralizing Antibody (NAb) in Participants With a Positive ADA by Visit
Time Frame: Day 1 up to Day 169
Population: mITT population. Only participants with a positive ADA status were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab-Pfizer | Rituximab-EU | Rituximab-US
Number analyzed (Participants) | 35 | 39 | 34
Percentage of participants | 0.0 | 0.0 | 0.0

18. Secondary Outcome: Change From Baseline in Disease Activity Score Based on 28-Joint Count and C-Reactive Protein (DAS28-CRP)
Description: DAS28-CRP was calculated from the swollen joint count and tender joint count using the 28 joints count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-CRP less than or equal to (≤)3.2 implied low disease activity, DAS28-CRP greater than (>)3.2 to ≤5.1 implied moderate to high disease activity, and DAS28-CRP less than (<)2.6 implied remission.
Time Frame: Baseline and Weeks 3, 5, 9, 13, 17, 21 and 25
Population: mITT population. "Number Analyzed" = participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rituximab-Pfizer | Rituximab-EU | Rituximab-US
Number analyzed (Participants) | 73 | 74 | 73
Units on a scale
  Baseline | 5.6862 (0.85109) | 5.7928 (0.9503) | 6.2221 (0.88162)
  Change at Week 3: number analyzed (Participants) | 69 | 74 | 69
  Change at Week 3 | -0.9 (1.01) | -0.8 (1.13) | -1.1 (1.02)
  Change at Week 5: number analyzed (Participants) | 71 | 71 | 67
  Change at Week 5 | -1.4 (1.17) | -1.4 (1.06) | -1.6 (1.20)
  Change at Week 9: number analyzed (Participants) | 68 | 73 | 70
  Change at Week 9 | -1.7 (1.29) | -1.8 (1.3) | -2.1 (1.37)
  Change at Week 13: number analyzed (Participants) | 67 | 72 | 67
  Change at Week 13 | -2.0 (1.43) | -2.1 (1.33) | -2.3 (1.34)
  Change at Week 17: number analyzed (Participants) | 66 | 71 | 67
  Change at Week 17 | -2.0 (1.32) | -2.1 (1.39) | -2.4 (1.35)
  Change at Week 21: number analyzed (Participants) | 60 | 65 | 59
  Change at Week 21 | -2.0 (1.28) | -1.9 (1.33) | -2.6 (1.35)
  Change at Week 25: number analyzed (Participants) | 50 | 58 | 55
  Change at Week 25 | -1.7 (1.25) | -2.0 (1.30) | -2.5 (1.30)

19. Secondary Outcome: Percent Change From Baseline in DAS28-CRP by Visit
Description: as for outcome 18
Time Frame: Baseline and Weeks 3, 5, 9, 13, 17, 21 and 25
Population: mITT population. "Number Analyzed" = participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Rituximab-Pfizer | Rituximab-EU | Rituximab-US
Number analyzed (Participants) | 73 | 74 | 73
Percent change
  Week 3: number analyzed (Participants) | 69 | 74 | 69
  Week 3 | -16.1 (19.08) | -13.6 (20.41) | -18.6 (17.63)
  Week 5: number analyzed (Participants) | 71 | 71 | 67
  Week 5 | -25.4 (20.74) | -24.0 (18.22) | -26.0 (21.88)
  Week 9: number analyzed (Participants) | 68 | 73 | 70
  Week 9 | -31.2 (22.31) | -31.0 (21.92) | -34.2 (22.97)
  Week 13: number analyzed (Participants) | 67 | 72 | 67
  Week 13 | -34.7 (24.0) | -36.9 (22.1) | -37.4 (21.42)
  Week 17: number analyzed (Participants) | 66 | 71 | 67
  Week 17 | -34.9 (22.65) | -35.4 (23.28) | -39.1 (21.35)
  Week 21: number analyzed (Participants) | 60 | 65 | 59
  Week 21 | -35.5 (21.99) | -33.4 (22.56) | -43.2 (21.39)
  Week 25: number analyzed (Participants) | 50 | 58 | 55
  Week 25 | -31.1 (22.72) | -34.6 (22.25) | -40.0 (20.55)

20. Secondary Outcome: Percentage of Participants With Good European League Against Rheumatism (EULAR) Response Based on Disease Activity Score Based on 28-Joint Count (DAS28) by Visit
Description: The DAS28-based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders: change from baseline >1.2 with DAS28 ≤3.2; moderate responders: change from baseline >1.2 with DAS28 >3.2 to ≤5.1 or change from baseline >0.6 to ≤1.2 with DAS28 ≤5.1; non-responders: change from baseline ≤0.6, or change from baseline >0.6 and ≤1.2 with DAS28 >5.1.
Time Frame: Weeks 3, 5, 9, 13, 17, 21 and 25
Population: mITT population. "Number Analyzed" = participants evaluable at specified time points.
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab-Pfizer | Rituximab-EU | Rituximab-US
Number analyzed (Participants) | 73 | 74 | 73
Percentage of participants
  Week 3: number analyzed (Participants) | 69 | 74 | 69
  Week 3 | 14.5 | 10.8 | 8.7
  Week 5: number analyzed (Participants) | 71 | 71 | 67
  Week 5 | 22.5 | 22.5 | 19.4
  Week 9: number analyzed (Participants) | 68 | 73 | 70
  Week 9 | 30.9 | 31.5 | 25.7
  Week 13: number analyzed (Participants) | 67 | 72 | 67
  Week 13 | 41.8 | 44.4 | 32.8
  Week 17: number analyzed (Participants) | 66 | 71 | 67
  Week 17 | 36.4 | 38.0 | 32.8
  Week 21: number analyzed (Participants) | 60 | 65 | 59
  Week 21 | 35.0 | 35.4 | 47.5
  Week 25: number analyzed (Participants) | 50 | 58 | 55
  Week 25 | 30.0 | 36.2 | 41.8

21. Secondary Outcome: Percentage of Participants With Moderate EULAR Response Based on Disease Activity Score Based on DAS28 by Visit
Description: as for outcome 20
Time Frame: Weeks 3, 5, 9, 13, 17, 21 and 25
Population: mITT population. "Number Analyzed" = participants evaluable at specified time points.
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab-Pfizer | Rituximab-EU | Rituximab-US
Number analyzed (Participants) | 73 | 74 | 73
Percentage of participants
  Week 3: number analyzed (Participants) | 69 | 74 | 69
  Week 3 | 33.3 | 35.1 | 42.0
  Week 5: number analyzed (Participants) | 71 | 71 | 67
  Week 5 | 47.9 | 39.4 | 43.3
  Week 9: number analyzed (Participants) | 68 | 73 | 70
  Week 9 | 45.6 | 43.8 | 54.3
  Week 13: number analyzed (Participants) | 67 | 72 | 67
  Week 13 | 38.8 | 37.5 | 44.8
  Week 17: number analyzed (Participants) | 66 | 71 | 67
  Week 17 | 45.5 | 39.4 | 53.7
  Week 21: number analyzed (Participants) | 60 | 65 | 59
  Week 21 | 51.7 | 46.2 | 39.0
  Week 25: number analyzed (Participants) | 50 | 58 | 55
  Week 25 | 50.0 | 46.6 | 43.6

22. Secondary Outcome: Percentage of Participants With No EULAR Response Based on DAS28 by Visit
Description: as for outcome 20
Time Frame: Weeks 3, 5, 9, 13, 17, 21 and 25
Population: mITT population. "Number Analyzed" = participants evaluable at specified time points.
Measure: Number; unit: Percentage of Participants
Arm/Group | Rituximab-Pfizer | Rituximab-EU | Rituximab-US
Number analyzed (Participants) | 73 | 74 | 73
Percentage of Participants
  Week 3: number analyzed (Participants) | 69 | 74 | 69
  Week 3 | 52.2 | 54.1 | 49.3
  Week 5: number analyzed (Participants) | 71 | 71 | 67
  Week 5 | 29.6 | 38.0 | 37.3
  Week 9: number analyzed (Participants) | 68 | 73 | 70
  Week 9 | 23.5 | 24.7 | 20.0
  Week 13: number analyzed (Participants) | 67 | 72 | 67
  Week 13 | 19.4 | 18.1 | 22.4
  Week 17: number analyzed (Participants) | 66 | 71 | 67
  Week 17 | 18.2 | 22.5 | 13.4
  Week 21: number analyzed (Participants) | 60 | 65 | 59
  Week 21 | 13.3 | 18.5 | 13.6
  Week 25: number analyzed (Participants) | 50 | 58 | 55
  Week 25 | 20.0 | 17.2 | 14.5

23. Secondary Outcome: Percentage of Participants With Low Disease Activity Score (DAS <=3.2) by Visit
Description: DAS28-CRP was calculated from the swollen joint count and tender joint count using the 28 joints count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-CRP ≤3.2 implied low disease activity. p-value of 9999 indicates p-value is not applicable.
Time Frame: Weeks 3, 5, 9, 13, 17, 21 and 25
Population: mITT population. "Number Analyzed" = participants evaluable at specified time points.
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab-Pfizer | Rituximab-EU | Rituximab-US
Number analyzed (Participants) | 73 | 74 | 73
Percentage of participants
  Week 3: number analyzed (Participants) | 69 | 74 | 69
  Week 3 | 14.5 | 10.8 | 10.1
  Week 5: number analyzed (Participants) | 71 | 71 | 67
  Week 5 | 23.9 | 25.4 | 19.4
  Week 9: number analyzed (Participants) | 68 | 73 | 70
  Week 9 | 30.9 | 32.9 | 25.7
  Week 13: number analyzed (Participants) | 67 | 72 | 67
  Week 13 | 41.8 | 44.4 | 32.8
  Week 17: number analyzed (Participants) | 66 | 71 | 67
  Week 17 | 36.4 | 38.0 | 32.8
  Week 21: number analyzed (Participants) | 60 | 65 | 59
  Week 21 | 35.0 | 36.9 | 47.5
  Week 25: number analyzed (Participants) | 50 | 58 | 55
  Week 25 | 32.0 | 37.9 | 41.8
Statistical Analysis 1: Comparison: Rituximab-Pfizer vs Rituximab-EU; Statistical analysis of rituximab-EU versus rituximab-Pfizer at Week 3; Test type: Superiority; Risk Ratio (RR) = 0.75, 95% CI 2-sided [0.31 to 1.78] — Rituximab-EU is the numerator
Statistical Analysis 2: Comparison: Rituximab-Pfizer vs Rituximab-EU; Statistical analysis of rituximab-EU versus rituximab-Pfizer at Week 5; Test type: Superiority; Risk Ratio (RR) = 1.06, 95% CI 2-sided [0.60 to 1.88] — Rituximab-EU is the numerator
Statistical Analysis 3: Comparison: Rituximab-Pfizer vs Rituximab-EU; Statistical analysis of rituximab-EU versus rituximab-Pfizer at Week 9; Test type: Superiority; Risk Ratio (RR) = 1.06, 95% CI 2-sided [0.66 to 1.73] — Rituximab-EU is the numerator
Statistical Analysis 4: Comparison: Rituximab-Pfizer vs Rituximab-EU; Statistical analysis of rituximab-EU versus rituximab-Pfizer at Week 13; Test type: Superiority; Risk Ratio (RR) = 1.06, 95% CI 2-sided [0.73 to 1.56] — Rituximab-EU is the numerator
Statistical Analysis 5: Comparison: Rituximab-Pfizer vs Rituximab-EU; Statistical analysis of rituximab-EU versus rituximab-Pfizer at Week 17; Test type: Superiority; Risk Ratio (RR) = 1.05, 95% CI 2-sided [0.68 to 1.62] — Rituximab-EU is the numerator
Statistical Analysis 6: Comparison: Rituximab-Pfizer vs Rituximab-EU; Statistical analysis of rituximab-EU versus rituximab-Pfizer at Week 21; Test type: Superiority; Risk Ratio (RR) = 1.05, 95% CI 2-sided [0.66 to 1.69] — Rituximab-EU is the numerator
Statistical Analysis 7: Comparison: Rituximab-Pfizer vs Rituximab-EU; Statistical analysis of rituximab-EU versus rituximab-Pfizer at Week 25 (EOT); Test type: Superiority; Risk Ratio (RR) = 1.19, 95% CI 2-sided [0.70 to 2.00] — Rituximab-EU is the numerator
Statistical Analysis 8: Comparison: Rituximab-Pfizer vs Rituximab-US; Statistical analysis of rituximab-US versus rituximab-Pfizer at Week 3; Test type: Superiority; Risk Ratio (RR) = 0.70, 95% CI 2-sided [0.28 to 1.73] — Rituximab-US is the numerator
Statistical Analysis 9: Comparison: Rituximab-Pfizer vs Rituximab-US; Statistical analysis of rituximab-US versus rituximab-Pfizer at Week 5; Test type: Superiority; Risk Ratio (RR) = 0.81, 95% CI 2-sided [0.43 to 1.54] — Rituximab-US is the numerator
Statistical Analysis 10: Comparison: Rituximab-Pfizer vs Rituximab-US; Statistical analysis of rituximab-US versus rituximab-Pfizer at Week 9; Test type: Superiority; Risk Ratio (RR) = 0.83, 95% CI 2-sided [0.49 to 1.42] — Rituximab-US is the numerator
Statistical Analysis 11: Comparison: Rituximab-Pfizer vs Rituximab-US; Statistical analysis of rituximab-US versus rituximab-Pfizer at Week 13; Test type: Superiority; Risk Ratio (RR) = 0.79, 95% CI 2-sided [0.50 to 1.22] — Rituximab-US is the numerator
Statistical Analysis 12: Comparison: Rituximab-Pfizer vs Rituximab-US; Statistical analysis of rituximab-US versus rituximab-Pfizer at Week 17; Test type: Superiority; Risk Ratio (RR) = 0.90, 95% CI 2-sided [0.57 to 1.44] — Rituximab-US is the numerator
Statistical Analysis 13: Comparison: Rituximab-Pfizer vs Rituximab-US; Statistical analysis of rituximab-US versus rituximab-Pfizer at Week 21; Test type: Superiority; Risk Ratio (RR) = 1.36, 95% CI 2-sided [0.88 to 2.10] — Rituximab-US is the numerator
Statistical Analysis 14: Comparison: Rituximab-Pfizer vs Rituximab-US; Statistical analysis of rituximab-US versus rituximab-Pfizer at Week 25 (EOT); Test type: Superiority; Risk Ratio (RR) = 1.31, 95% CI 2-sided [0.78 to 2.18] — Rituximab-US is the numerator
Statistical Analysis 15: Comparison: Rituximab-EU vs Rituximab-US; Statistical analysis of rituximab-US versus rituximab-EU at Week 3; Test type: Superiority; Risk Ratio (RR) = 0.94, 95% CI 2-sided [0.36 to 2.45] — Rituximab-US is the numerator
Statistical Analysis 16: Comparison: Rituximab-EU vs Rituximab-US; Statistical analysis of rituximab-US versus rituximab-EU at Week 5; Test type: Superiority; Risk Ratio (RR) = 0.77, 95% CI 2-sided [0.41 to 1.44] — Rituximab-US is the numerator
Statistical Analysis 17: Comparison: Rituximab-EU vs Rituximab-US; Statistical analysis of rituximab-US versus rituximab-EU at Week 9; Test type: Superiority; Risk Ratio (RR) = 0.78, 95% CI 2-sided [0.47 to 1.31] — Rituximab-US is the numerator
Statistical Analysis 18: Comparison: Rituximab-EU vs Rituximab-US; Statistical analysis of rituximab-US versus rituximab-EU at Week 13; Test type: Superiority; Risk Ratio (RR) = 0.74, 95% CI 2-sided [0.48 to 1.13] — Rituximab-US is the numerator
Statistical Analysis 19: Comparison: Rituximab-EU vs Rituximab-US; Statistical analysis of rituximab-US versus rituximab-EU at Week 17; Test type: Superiority; Risk Ratio (RR) = 0.86, 95% CI 2-sided [0.55 to 1.36] — Rituximab-US is the numerator
Statistical Analysis 20: Comparison: Rituximab-EU vs Rituximab-US; Statistical analysis of rituximab-US versus rituximab-EU at Week 21; Test type: Superiority; Risk Ratio (RR) = 1.29, 95% CI 2-sided [0.85 to 1.95] — Rituximab-US is the numerator
Statistical Analysis 21: Comparison: Rituximab-EU vs Rituximab-US; Statistical analysis of rituximab-US versus rituximab-EU at Week 25 (EOT); Test type: Superiority; Risk Ratio (RR) = 1.10, 95% CI 2-sided [0.70 to 1.73] — Rituximab-US is the numerator

24. Secondary Outcome: Percentage of Participants With DAS Remission (DAS <2.6) by Visit
Description: DAS28-CRP was calculated from the swollen joint count and tender joint count using the 28 joints count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-CRP <2.6 implied remission. p-value of 9999 indicates p-value is not applicable.
Time Frame: Weeks 3, 5, 9, 13, 17, 21 and 25
Population: mITT population. "Number Analyzed" = participants evaluable at specified time points.
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab-Pfizer | Rituximab-EU | Rituximab-US
Number analyzed (Participants) | 73 | 74 | 73
Percentage of participants
  Week 3: number analyzed (Participants) | 69 | 74 | 69
  Week 3 | 8.7 | 4.1 | 7.2
  Week 5: number analyzed (Participants) | 71 | 71 | 67
  Week 5 | 16.9 | 8.5 | 11.9
  Week 9: number analyzed (Participants) | 68 | 73 | 70
  Week 9 | 26.5 | 20.5 | 20.0
  Week 13: number analyzed (Participants) | 67 | 72 | 67
  Week 13 | 28.4 | 29.2 | 25.4
  Week 17: number analyzed (Participants) | 66 | 71 | 67
  Week 17 | 25.8 | 25.4 | 23.9
  Week 21: number analyzed (Participants) | 60 | 65 | 59
  Week 21 | 25.0 | 16.9 | 30.5
  Week 25: number analyzed (Participants) | 50 | 58 | 55
  Week 25 | 28.0 | 24.1 | 23.6
Statistical Analysis 1: Comparison: Rituximab-Pfizer vs Rituximab-EU; Statistical analysis of rituximab-EU versus rituximab-Pfizer at Week 3; Test type: Superiority; Risk Ratio (RR) = 0.47, 95% CI 2-sided [0.12 to 1.79] — Rituximab-EU is the numerator
Statistical Analysis 2: Comparison: Rituximab-Pfizer vs Rituximab-EU; Statistical analysis of rituximab-EU versus rituximab-Pfizer at Week 5; Test type: Superiority; Risk Ratio (RR) = 0.50, 95% CI 2-sided [0.20 to 1.26] — Rituximab-EU is the numerator
Statistical Analysis 3: Comparison: Rituximab-Pfizer vs Rituximab-EU; Statistical analysis of rituximab-EU versus rituximab-Pfizer at Week 9; Test type: Superiority; Risk Ratio (RR) = 0.78, 95% CI 2-sided [0.43 to 1.41] — Rituximab-EU is the numerator
Statistical Analysis 4: Comparison: Rituximab-Pfizer vs Rituximab-EU; Statistical analysis of rituximab-EU versus rituximab-Pfizer at Week 13; Test type: Superiority; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.61 to 1.74] — Rituximab-EU is the numerator
Statistical Analysis 5: Comparison: Rituximab-Pfizer vs Rituximab-EU; Statistical analysis of rituximab-EU versus rituximab-Pfizer at Week 17; Test type: Superiority; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.56 to 1.74] — Rituximab-EU is the numerator
Statistical Analysis 6: Comparison: Rituximab-Pfizer vs Rituximab-EU; Statistical analysis of rituximab-EU versus rituximab-Pfizer at Week 21; Test type: Superiority; Risk Ratio (RR) = 0.68, 95% CI 2-sided [0.34 to 1.36] — Rituximab-EU is the numerator
Statistical Analysis 7: Comparison: Rituximab-Pfizer vs Rituximab-EU; Statistical analysis of rituximab-EU versus rituximab-Pfizer at Week 25 (EOT); Test type: Superiority; Risk Ratio (RR) = 0.86, 95% CI 2-sided [0.46 to 1.63] — Rituximab-EU is the numerator
Statistical Analysis 8: Comparison: Rituximab-Pfizer vs Rituximab-US; Statistical analysis of rituximab-US versus rituximab-Pfizer at Week 3; Test type: Superiority; Risk Ratio (RR) = 0.83, 95% CI 2-sided [0.27 to 2.60] — Rituximab-US is the numerator
Statistical Analysis 9: Comparison: Rituximab-Pfizer vs Rituximab-US; Statistical analysis of rituximab-US versus rituximab-Pfizer at Week 5; Test type: Superiority; Risk Ratio (RR) = 0.71, 95% CI 2-sided [0.31 to 1.62] — Rituximab-US is the numerator
Statistical Analysis 10: Comparison: Rituximab-Pfizer vs Rituximab-US; Statistical analysis of rituximab-US versus rituximab-Pfizer at Week 9; Test type: Superiority; Risk Ratio (RR) = 0.76, 95% CI 2-sided [0.41 to 1.40] — Rituximab-US is the numerator
Statistical Analysis 11: Comparison: Rituximab-Pfizer vs Rituximab-US; Statistical analysis of rituximab-US versus rituximab-Pfizer at Week 13; Test type: Superiority; Risk Ratio (RR) = 0.89, 95% CI 2-sided [0.51 to 1.57] — Rituximab-US is the numerator
Statistical Analysis 12: Comparison: Rituximab-Pfizer vs Rituximab-US; Statistical analysis of rituximab-US versus rituximab-Pfizer at Week 17; Test type: Superiority; Risk Ratio (RR) = 0.93, 95% CI 2-sided [0.51 to 1.68] — Rituximab-US is the numerator
Statistical Analysis 13: Comparison: Rituximab-Pfizer vs Rituximab-US; Statistical analysis of rituximab-US versus rituximab-Pfizer at Week 21; Test type: Superiority; Risk Ratio (RR) = 1.22, 95% CI 2-sided [0.68 to 2.19] — Rituximab-US is the numerator
Statistical Analysis 14: Comparison: Rituximab-Pfizer vs Rituximab-US; Statistical analysis of rituximab-US versus rituximab-Pfizer at Week 25 (EOT); Test type: Superiority; Risk Ratio (RR) = 0.84, 95% CI 2-sided [0.44 to 1.62] — Rituximab-US is the numerator
Statistical Analysis 15: Comparison: Rituximab-EU vs Rituximab-US; Statistical analysis of rituximab-US versus rituximab-EU at Week 3; Test type: Superiority; Risk Ratio (RR) = 1.79, 95% CI 2-sided [0.44 to 7.20] — Rituximab-US is the numerator
Statistical Analysis 16: Comparison: Rituximab-EU vs Rituximab-US; Statistical analysis of rituximab-US versus rituximab-EU at Week 5; Test type: Superiority; Risk Ratio (RR) = 1.41, 95% CI 2-sided [0.52 to 3.86] — Rituximab-US is the numerator
Statistical Analysis 17: Comparison: Rituximab-EU vs Rituximab-US; Statistical analysis of rituximab-US versus rituximab-EU at Week 9; Test type: Superiority; Risk Ratio (RR) = 0.97, 95% CI 2-sided [0.51 to 1.87] — Rituximab-US is the numerator
Statistical Analysis 18: Comparison: Rituximab-EU vs Rituximab-US; Statistical analysis of rituximab-US versus rituximab-EU at Week 13; Test type: Superiority; Risk Ratio (RR) = 0.87, 95% CI 2-sided [0.50 to 1.50] — Rituximab-US is the numerator
Statistical Analysis 19: Comparison: Rituximab-EU vs Rituximab-US; Statistical analysis of rituximab-US versus rituximab-EU at Week 17; Test type: Superiority; Risk Ratio (RR) = 0.94, 95% CI 2-sided [0.52 to 1.69] — Rituximab-US is the numerator
Statistical Analysis 20: Comparison: Rituximab-EU vs Rituximab-US; Statistical analysis of rituximab-US versus rituximab-EU at Week 21; Test type: Superiority; Risk Ratio (RR) = 1.80, 95% CI 2-sided [0.93 to 3.50] — Rituximab-US is the numerator
Statistical Analysis 21: Comparison: Rituximab-EU vs Rituximab-US; Statistical analysis of rituximab-US versus rituximab-EU at Week 25 (EOT); Test type: Superiority; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.51 to 1.89] — Rituximab-US is the numerator

25. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) by Visit
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline, Week 3, 5, 9, 13, 17, 21 and 25
Population: mITT population. "Number Analyzed" = participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rituximab-Pfizer | Rituximab-EU | Rituximab-US
Number analyzed (Participants) | 73 | 74 | 73
Units on a scale
  Baseline | 1.6541 (0.57340) | 1.5929 (0.53597) | 1.7466 (0.62081)
  Change at Week 3: number analyzed (Participants) | 70 | 74 | 70
  Change at Week 3 | -0.2 (0.39) | -0.2 (0.34) | -0.2 (0.33)
  Change at Week 5: number analyzed (Participants) | 72 | 70 | 68
  Change at Week 5 | -0.3 (0.39) | -0.3 (0.45) | -0.3 (0.43)
  Change at Week 9: number analyzed (Participants) | 68 | 73 | 70
  Change at Week 9 | -0.4 (0.47) | -0.5 (0.50) | -0.5 (0.54)
  Change at Week 13: number analyzed (Participants) | 67 | 72 | 68
  Change at Week 13 | -0.4 (0.55) | -0.6 (0.56) | -0.5 (0.52)
  Change at Week 17: number analyzed (Participants) | 66 | 71 | 67
  Change at Week 17 | -0.3 (0.49) | -0.6 (0.58) | -0.5 (0.55)
  Change at Week 21: number analyzed (Participants) | 63 | 70 | 64
  Change at Week 21 | -0.4 (0.53) | -0.6 (0.58) | -0.6 (0.61)
  Change at Week 25: number analyzed (Participants) | 52 | 59 | 55
  Change at Week 25 | -0.4 (0.49) | -0.5 (0.63) | -0.6 (0.57)

26. Secondary Outcome: Percent Change From Baseline in HAQ-DI Score by Visit
Description: as for outcome 25
Time Frame: Baseline, Week 3, 5, 9, 13, 17, 21 and 25
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Rituximab-Pfizer | Rituximab-EU | Rituximab-US
Number analyzed (Participants) | 72 | 74 | 73
Percentage change
  Week 3: number analyzed (Participants) | 70 | 74 | 70
  Week 3 | -10.4 (37.27) | -13.2 (26.03) | -9.0 (25.68)
  Week 5: number analyzed (Participants) | 72 | 70 | 68
  Week 5 | -15.1 (40.00) | -23.5 (30.45) | -14.8 (43.82)
  Week 9: number analyzed (Participants) | 68 | 73 | 70
  Week 9 | -22.4 (35.96) | -31.7 (34.64) | -24.5 (35.51)
  Week 13: number analyzed (Participants) | 67 | 72 | 68
  Week 13 | -14.6 (50.35) | -39.5 (37.46) | -30.7 (31.91)
  Week 17: number analyzed (Participants) | 66 | 71 | 67
  Week 17 | -16.9 (48.95) | -39.1 (38.85) | -28.8 (36.43)
  Week 21: number analyzed (Participants) | 63 | 70 | 64
  Week 21 | -21.0 (48.04) | -39.2 (38.34) | -33.5 (35.18)
  Week 25: number analyzed (Participants) | 52 | 59 | 55
  Week 25 | -17.7 (54.01) | -37.1 (41.18) | -38.4 (34.60)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for 28 days after the last administration of study drug or, in the case of incomplete B-cell count recovery, for up to 1 year after Study Day 1.
Description: The same event may appear as both an AE and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or 1 participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Rituximab-Pfizer | Rituximab-EU | Rituximab-US
Serious Adverse Events (participants affected / at risk) | 5/73 | 1/74 | 4/73
Other Adverse Events (participants affected / at risk) | 49/73 | 40/74 | 45/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab-Pfizer (N=73) | Rituximab-EU (N=74) | Rituximab-US (N=73)
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab-Pfizer (N=73) | Rituximab-EU (N=74) | Rituximab-US (N=73)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 5 | 5
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 4 | 2 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1
Venous insufficiency (Vascular disorders) | 0 | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 0
Ear disorder (Ear and labyrinth disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Ear pruritus (Ear and labyrinth disorders) | 2 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 1
Abnormal sensation in eye (Eye disorders) | 0 | 1 | 0
Blepharitis (Eye disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0
Eye haemorrhage (Eye disorders) | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 1
Eyelid pain (Eye disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 2
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 1
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 4
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Tongue ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Adverse drug reaction (General disorders) | 0 | 0 | 1
Asthenia (General disorders) | 3 | 0 | 0
Chest discomfort (General disorders) | 1 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 5 | 1 | 1
Inflammation (General disorders) | 1 | 0 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 1
Local swelling (General disorders) | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Extrasystoles (Cardiac disorders) | 1 | 0 | 0
Tachycardia paroxysmal (Cardiac disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 3 | 2 | 4
Cellulitis (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 1 | 1 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Infected bites (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 2 | 1 | 2
Nasopharyngitis (Infections and infestations) | 3 | 1 | 3
Oral herpes (Infections and infestations) | 0 | 0 | 1
Otitis externa (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 1 | 0
Sinusitis (Infections and infestations) | 3 | 6 | 2
Tooth abscess (Infections and infestations) | 1 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 7 | 5 | 4
Urinary tract infection (Infections and infestations) | 1 | 0 | 2
Viral infection (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 2
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Underdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Bilirubin conjugated increased (Investigations) | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Blood calcium increased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 1
Blood glucose increased (Investigations) | 1 | 0 | 0
Blood potassium decreased (Investigations) | 1 | 0 | 0
Blood pressure decreased (Investigations) | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 2 | 0
Blood urea increased (Investigations) | 0 | 1 | 1
Haematocrit decreased (Investigations) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Renal pain (Renal and urinary disorders) | 0 | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 2
Headache (Nervous system disorders) | 3 | 2 | 4
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 1 | 1 | 0
Migraine (Nervous system disorders) | 1 | 0 | 1
Neuralgia (Nervous system disorders) | 2 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 2 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 3
Depression (Psychiatric disorders) | 1 | 1 | 3
Insomnia (Psychiatric disorders) | 1 | 2 | 3
Mood swings (Psychiatric disorders) | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Campbell de Morgan spots (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less